CLINICAL TRIAL: NCT03574766
Title: Meditation for NICU Moms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Katherine Massa, MD, Maternal Fetal Medicine Fellow, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29082
Record Dates: First submitted 2018-05-10; First posted 2018-07-02 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Breast Feeding; Premature Birth; Stress; Depression, Postpartum; Anxiety; Self Efficacy; Behavior, Maternal; Insufficient Lactation
MeSH Terms: conditions — Breast Feeding; Premature Birth; Depression, Postpartum; Anxiety Disorders; Behavior; Lactation Disorders | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation Group (Experimental): Twenty minutes of daily meditation for 7 days. Routine lactation support.
  Interventions: Behavioral: Meditation
- Control Group (No Intervention): Routine lactation support.

INTERVENTIONS:
Behavioral: Meditation — Daily meditation
  Other Names: Expectful App meditation
  Arms: Meditation Group

SUMMARY:
This project explores whether meditation increases breastmilk supply in mothers who are pumping milk for infants in the NICU. Mothers will be randomly assigned to daily meditation while pumping using an app designed for meditation for new mothers, and their breastmilk volume will be measured after one week of meditation versus a control group with measurements at the same time points. Investigators will also determine whether mediation improves breastfeeding confidence and reduces stress, anxiety and depression symptoms in these mothers. Finally investigators will examine the effect on salivary cortisol levels.

ELIGIBILITY:
Inclusion Criteria:

* 1) Mothers of all ages, including emancipated minors will be included 2) Gestational age at birth of 24 completed weeks to 32 weeks 6 days 3) Mothers of infants admitted to St. Mary's NICU or with transfer or anticipated transfer to Cardinal Glennon NICU 4) Mothers who intend to provide breastmilk to infants for at least 1 month. 5) Recruitment within 24 hours of time of delivery in order to allow for beginning of 24 hour milk collection at 24 hours post delivery

Exclusion Criteria:

* 1) Mothers of infants expected to be nippling at the breast in less than 10 days 2) Infants for whom discharge is anticipated in less than 10 days 3) Participation in another interventional study at Screening or who plan to participate in another interventional study during the study period 4) Hearing loss that would preclude participation in meditation recordings 5) Inability to come for a midday (between 11am -3pm) visit on day of life #10. 6) Inability or unwillingness to perform the study procedures.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
24 hour breast milk volume | Post-Intervention/Infant Day of Life #9
  24 hours volume of pumped milk after 7 days of daily meditation collected versus change in pumped milk volume among mothers in a control group

SECONDARY OUTCOMES:
Perceived Stress Score:NICU | Post-intervention/Infant Day of Life # 10
  Comparison in the change in scores of Perceived Stress Score: NICU between Meditation Group and Control Group.
  This is a 26-question written questionnaire that evaluates parental stress in relation to the experiences of having an infant in the NICU.
  Subscales are the following:
  Sights and Sounds (5 questions) Baby looks and behaves and Treatments (14 questions) Relationship/Parental Role (7 questions)
  Question responses are on a scale of NA, 1, 2, 3, 4, 5
  Total scores range from NA to 130.A higher score on the scale indicates higher stress.
State-Trait Anxiety Inventory (STAI) | Post-intervention/Infant Day of Life # 10
  Comparison in the change in scores of State-Trait Anxiety Inventory between Meditation Group and Control Group.
  This is a 40-question written questionnaire that evaluates anxiety symptoms. Comparison of Baseline/Infant Day of Life #1 to Post-intervention/Infant Day of Life # 10.
  Question responses are on a scale of 1-4
  Total score ranges from 40-160. Scores are weighted using a scoring tool. A higher score is higher anxiety.
Edinburgh Postnatal Depression Scale (EPDS) | Post-intervention/Infant Day of Life # 10
  Comparison in the change in scores of Edinburgh Postnatal Depression Scale between the Meditation Group and Control Group
  This is a 10-question written questionnaire that evaluates depression symptoms. Maximum Score: 30 Possible Depression: 10 or greater Score 13 or greater = likely to be suffering from a depressive illness of varying severity Always look at Item 10 (suicidal thoughts)
Breastfeeding Self-Efficacy Scale-short Form with additional questions for critically ill infants | Post-intervention/Infant Day of Life # 10
  Comparison of scores Breastfeeding Self-Efficacy Scale-short Form with additional questions for critically ill infants between the Meditation Group and Control Group
  This is a 18-question questionnaire that evaluates breastfeeding self-efficacy in breastfeeding mothers of infants in the NICU. This scale will be used to assess breastfeeding self-efficacy.
  Question responses are on a scale of 1-5. Total score ranges from 18- 9. A higher score indicates higher confidence.
Salivary Cortisol - Hormonal regulation of breastfeeding and stress response | Infant Day of Life #9
  Diurnal salivary cortisol slope and cortisol awakening response with meditation versus without meditation.
Serum Cortisol hormone -Hormonal regulation of breastfeeding and stress response | Infant Day of Life #10
  Cortisol hormone during milk expression with meditation versus without meditation.
Serum Adrenocorticotrophic hormone -Hormonal regulation of breastfeeding and stress response | Infant Day of Life #10
  Adrenocorticotrophic hormone during milk expression with meditation versus without meditation.
Serum Catecholamines -Hormonal regulation of breastfeeding and stress response | Infant Day of Life #10
  Catecholamines during milk expression with meditation versus without meditation.
Serum Dihydroepiandosterone - Hormonal regulation of breastfeeding and stress response | Infant Day of Life #10
  Dihydroepiandosterone during milk expression with meditation versus without meditation.
Number of skin-to-skin episodes -Lactation promoting behaviors | Day of Life #1 through Infant Day of Life #9
  Number of skin-to-skin episodes between Infant Day of Life #1 and Infant Day of Life #9 recorded in daily diary
Use of hand expression - Lactation promoting behaviors | Infant Day of Life #9
  Use of hand expression with breastmilk pumping
Pumping episodes -Lactation promoting behaviors | Post-Intervention/Infant Day of Life #9
  number of reported pumping episodes reported in 24-hour milk collection log
Supplementation of infant feeding with formula or donor human breastmilk | 4 weeks post-partum
  Supplementation of infant feeding with formula or donor human breastmilk
Sustained breastfeeding at 4 weeks postpartum | 4 weeks postpartum
  Sustained breastfeeding at 4 weeks postpartum, supplementation feeding with formula or donor milk at 2 and 4 weeks postpartum
  Mother is asked if she is still providing breast milk (No/Yes) and if Baby is fed exclusively with mother's breastmilk (No/Yes) at 2 and 4 weeks postpartum
Duration of meditation | 4 weeks postpartum
  Duration of meditation at 4 weeks postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- St. Mary's Hospital, Richmond Heights, Missouri, United States